CLINICAL TRIAL: NCT04278768
Title: A Phase 1/2A, Open Label Dose Escalation and Expansion Study of Orally Administered CA-4948 as a Monotherapy in Patients With Acute Myelogenous Leukemia or Myelodysplastic Syndrome
Brief Title: Dose Escalation/ Expansion Study of CA-4948 as Monotherapy in Patients With Acute Myelogenous Leukemia (AML) or Myelodysplastic Syndrome (MDS)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Curis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CA-4948-102
Record Dates: First submitted 2020-02-10; First posted 2020-02-20 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Acute Myelogenous Leukemia; Myelodysplastic Syndrome
Keywords: Acute Myelogenous Leukemia; Myelodysplastic Syndrome; AML; MDS; Interleukin-1 receptor-associated kinase 4 (IRAK4); FLT3-ITD or TKD mutant; FLT3 Wild Type (WT); Relapse/refractory to hypomethylating agent (HMA); spliceosome mutation; SF3B1; U2AF1; Serine/arginine-rich splicing factor 2 (SRSF2); Zinc finger CCCH-type, RNA binding motif and serine/arginine rich 2 (ZRSR2); higher-risk MDS; failing prior treatment; R/R AML or relapse/refractory AML; R/R hrMDS or relapse/refractory hrMDS; FLT3 mutation; FLT3 inhibitor
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Hereditary Sensory and Autonomic Neuropathies; Recurrence | interventions — CA-4948; venetoclax

STUDY DESIGN:
Intervention Model Description: Phase 1 and 1b follow a 3 + 3 design where 3 patients will be enrolled at the starting dose level. If none of the first 3 patients experience a DLT during the 1st cycle, patients may be enrolled into the next higher dose level. If 1 patient out of the first 3 experiences a DLT, the dose level may be expanded with an additional 3 patients. If 2 or 3 patients out of the first six experience a DLT, this will be considered a DLT rate above the max tolerated dose (> 33%), and additional enrollment will proceed at a lower dose level. The Phase 2a Dose Expansion will be enrolled after the RP2D is determined from Phase 1. It will be in 3 Cohorts of patients: (1) R/R AML with FTLT-3 mutation who have been previously treated with a FLT3 inhibitor; (2) R/R AML with spliceosome mutations of SF3B1 or U2AF1; and (3) R/R hrMDS (IPSS-R >3.5) with spliceosome mutations of SF3B1 or U2AF1; AND all patients have ≤ 2 lines of prior systemic anti-cancer therapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Emavusertib (CA-4948) dose escalation (Experimental): Patients receive emavusertib monotherapy BID daily. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Emavusertib
- Emavusertib dose escalation + Venetoclax (Experimental): The starting dose for emavusertib will be 200 mg BID for 21 days of a 28-day Cycle. Anticipated emavusertib doses will be 200 and 300 mg BID. Venetoclax will be administered at 100 mg orally (Day 1) per the product label at the same time each day with a ramp up over 3 days to 400 mg for 21days of a 28-day Cycle. Second and subsequent cycles start with target dose level.
  Interventions: Drug: Venetoclax; Drug: Emavusertib
- Emavusertib monotherapy dose expansion (Experimental): The Expansion phase will begin once the RP2D from Phase 1 Dose Escalation phase has been identified. There will be 3 Cohorts and patients will be assigned to each Cohort based on baseline disease.
  Interventions: Drug: Emavusertib

INTERVENTIONS:
Drug: Emavusertib — Emavusertib is formulated as a tablet for oral administration for BID dosing in consecutive 28-day cycles. Emavusertib is a novel small molecule inhibitor of interleukin-1 receptor-associated kinase 4 (IRAK4). IRAK4 kinase plays an essential role in toll-like receptor (TLR) and interleukin-1 receptor (IL-1R) signaling pathways and these pathways are frequently dysregulated in non-Hodgkin's lymphoma and AML/MDS malignancies.
  Other Names: CA-4948
  Arms: Emavusertib (CA-4948) dose escalation; Emavusertib monotherapy dose expansion
Drug: Venetoclax — Ventoclax is B-cell lymphoma-2 (BCL-2) inhibitor. Venetoclax will be administered at 100 mg orally (Day 1) per the product label at the same time each day with a ramp up over 3 days to 400 mg for 21days of a 28-day Cycle. Second and subsequent cycles start with target dose level.
  This arm of the study has been closed to enrollment.
  Arms: Emavusertib dose escalation + Venetoclax
Drug: Emavusertib — Emavusertib is formulated as a tablet for oral administration for BID dosing for 21 days (Days 1-21) of a 28-day Cycle.
  Other Names: CA-4948
  Arms: Emavusertib dose escalation + Venetoclax

SUMMARY:
This is a multicenter, open-label, Phase 1/2a dose escalation and expansion study of orally administered emavusertib (CA-4948) monotherapy in adult patients with AML or higher- risk Myelodysplastic Syndrome (hrMDS).

Patients enrolling in the Phase 1 dose escalation of the study must meet one of the following criteria prior to consenting to the study:

* Relapse/refractory (R/R) AML with FMS-like tyrosine kinase-3 (FLT3) mutations who have been previously treated with a FLT3 inhibitor
* R/R AML with spliceosome mutations of splicing factor 3B subunit 1 (SF3B1) or U2AF1
* R/R hrMDS with spliceosome mutations of SF3B1 or U2 small nuclear RNA auxiliary factor 1 (U2AF1)
* Number of pretreatments: 1 or 2

The Phase 2a Dose Expansion will be in 3 Cohorts of patients:

1. R/R AML with FLT3 mutations who have been previously treated with a FLT3 inhibitor;
2. R/R AML with spliceosome mutations of SF3B1 or U2AF1; and
3. R/R hrMDS (Revised International Prognostic Scoring System [IPSS-R] score > 3.5) with spliceosome mutations of SF3B1 or U2AF1.

All patients above have had ≤ 2 lines of prior systemic anticancer treatment. In previous versions of this protocol there was a Phase 1b portion of the study, in which patients with AML or hrMDS received CA-4948 in combination with venetoclax. This part of the study is no longer open for enrollment.

DETAILED DESCRIPTION:
The primary objective of the Phase 1 portion of the study is to determine the maximum tolerated dose (MTD) and Recommended Phase 2 Dose (RP2D) for emavusertib in monotherapy in patients with AML, intermediate-2, high risk, or every high risk MDS based on the safety and tolerability, dose-limiting toxicities (DLTs), and Pharmacokinetic (PK)/Pharmacodynamic (PD) findings.

The primary objective of the Phase 1b portion of the study is to determine MTD and RP2D for emavusertib in combination with azacitidine (AZA) in treatment naïve patients with hrMDS or in combination with venetoclax (VEN) in R/R patients with AML or hrMDS after first line treatment based on the safety and tolerability, DLTs and PK and pharmacodynamic findings. Note, this portion of the study is no longer enrolling patients.

The primary objective of the Phase 2a portion of the study (emavusertib monotherapy expansion) is to assess anti-cancer activity of CA-4948 at the RP2D in patients with R/R AML with FMS-like tyrosine kinase-3 (FLT3) mutations, or patients with R/R hrMDS or R/R AML with spliceosome mutations of SF3B1 or U2AF1.

Emavusertib is formulated as tablets for twice daily oral administration. Each treatment cycle will be 28 days in length and repeated in the absence of toxicity. Patients who tolerate emavusertib may continue to receive emavusertib until progression of disease, intolerable toxicity, lack of clinical benefit, withdrawal from the trial, or study termination.

The emavusertib starting dose level will be 200 milligrams (mg) twice daily (BID) which was determined to be safe, capable of achieving relevant levels of drug exposure as well as demonstrating signs of biologic activity and clinical efficacy in an ongoing study (Study CA-4948-101). For phase 1, emavusertib is taken daily for 28 days of a 28 day cycle. For Phase 1b, emavusertib is taken daily for 21 days of a 28 day cycle in combination with venetoclax.

Venetoclax will be administered at 100 mg orally (Day 1) per the product label at the same time each day with a ramp up over 3 days to 400 mg for 21 days of the 28-day Cycle. Second and subsequent cycles start with the target dose level.

In each of the Phase 1/1b cohorts, three patients with AML or MDS were enrolled at the designated dose. If none of the first 3 patients experience a DLT during the first cycle, patients may be enrolled into the next higher dose level. If 1 patient out of the first 3 experiences a DLT, the dose level may be expanded with an additional 3 patients. If 2 or 3 patients out of the first six experienced a DLT, this will be considered a DLT rate above the MTD (> 33%), and additional enrollment will proceed at a lower dose level. Any adverse reaction that led to dose reduction or discontinuation is considered a DLT unless the adverse reaction is clearly and solely related to disease.

The RP2D will be determined by the Clinical Safety Committee (CSC) in consultation with the Sponsor, considering all aspects of safety, tolerability, biologic activity, pharmacokinetics and preliminary efficacy in the trial population. The intent of the RP2D is to provide a dose and schedule that will maximize the opportunity for clinical benefit, while minimizing the risk of toxicity. The RP2D may be below the MTD. The CSC may request enrollment of additional patients at any previously-explored dose level in order to make an appropriate RP2D or MTD determination.

The expansion phase will begin once the RP2D from Phase 1 Dose Escalation phase has been identified. There will be 3 Cohorts and patients will be assigned to each Cohort based on baseline disease:

1. R/R AML with FLT3 mutations who have been previously treated with a FLT3 inhibitor; or
2. R/R AML with spliceosome mutations of SF3B1 or U2AF1; or
3. R/R hrMDS (IPSS-R score > 3.5) with spliceosome mutations of SF3B1 or U2AF1

All patients have had ≤ 2 lines of prior systemic anticancer treatment. This part of the study is no longer open for enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥18 years of age
2. Life expectancy of at least 3 months
3. Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤1
4. Cytomorphology based confirmed diagnosis of MDS or AML (as per World Health Organisation [WHO] 2016 classification) with the following characteristics.

   Phase 1 Dose Escalation (Monotherapy)

   • AML (primary or secondary, including treatment-related) after failing at least 1 standard treatment (may include chemotherapy, re induction therapy or stem cell transplantation).

   OR

   • Higher-risk R/R MDS that are considered resistant/refractory following at least 2 to 3 cycles of hypomethylating agent (HMA) or evidence of early progression

   Phase 2a Dose Expansion (Monotherapy)

   Patients with:
   * R/R AMLwith FLT3 mutations who have been previously treated with a FLT3 inhibitor
   * R/R AML with spliceosome mutations of SF3B1 or U2AF1
   * R/R hrMDS (IPSS-R score > 3.5) with spliceosome mutations of SF3B1 or U2AF1
   * Number of prior treatments: 1 or 2
5. Acceptable organ function at screening
6. Ability to swallow and retain oral medications
7. Negative serum pregnancy test in women of childbearing potential
8. Women of childbearing potential and men who partner with a woman of childbearing potential must agree to use highly effective contraceptive methods for the duration of the study and for 180 days after the last dose of emavusertib
9. Willing and able to provide written informed consent and comply with the requirements of the trial
10. Able to undergo serial bone marrow sampling and peripheral blood sampling

Exclusion Criteria:

1. Diagnosed with acute promyelocytic leukemia (APL, M3)
2. Has known active central nervous system (CNS) leukemia
3. Allogeneic hematopoietic stem cell transplant (Allo-HSCT) within 60 days of the first dose of emavusertib, or clinically significant graft-versus-host disease (GVHD) requiring ongoing up titration of immunosuppressive medications prior to start of emavusertib
4. Chronic myeloid leukemia (CML)
5. Any prior systemic anti-cancer treatment such as chemotherapy, immunomodulatory drug therapy, etc., received within 3 weeks (or 5 half-lives) prior to start of emavusertib.

   Localized radiation or surgical resection of skin cancers allowed.
6. Use of any investigational agent within 3 weeks or 5 half-lives, whichever is shorter, prior to start of emavusertib
7. Presence of an acute or chronic toxicity resulting from prior anti-cancer therapy, with the exception of alopecia that has not resolved to Grade ≤ 1 within 7 days prior to start of emavusertib.
8. Known allergy or hypersensitivity to any component of the formulation of emavusertib
9. Major surgery, other than diagnostic surgery, <28 days from the start of emavusertib; minor surgery <14 days from the start of emavusertib
10. Patients with active advanced malignant solid tumors
11. Known to be human immunodeficiency virus (HIV) positive or have an acquired immunodeficiency syndrome-related illness
12. Hepatitis B virus (HBV) deoxyribonucleic acid (DNA) positive or Hepatitis C virus (HCV) infection <6 months prior to start of emavusertib unless viral load is undetectable, or HCV with cirrhosis
13. Uncontrolled or severe cardiovascular disease including myocardial infarction or unstable angina within 6 months prior to CA-4948, New York Heart Association Class II or greater congestive heart failure, or left ventricular ejection fraction < 50% by echocardiogram or multi-gated acquisition scan, serious arrhythmias uncontrolled on treatment, clinically significant pericardial disease, cardiac amyloidosis, congenital long QT syndrome, or QTc with Fridericia's correction (QTcF) that is unmeasurable or > 450 milliseconds (msec) on Screening electrocardiogram (ECG)
14. Gastrointestinal disease or disorder that could interfere with the swallowing, oral absorption, or tolerance of emavusertib
15. Pregnant or lactating
16. Systemic fungal, bacterial, viral, or other infection that is not controlled
17. Any other severe, acute, or chronic medical, psychiatric or social condition, or laboratory abnormality that may increase the risk of trial participation or emavusertib administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Estimated)
Dates: Start 2020-07-06 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Determine Maximum Tolerated Dose (MTD) of emavusertib (CA-4948) monotherapy (Phase 1) | 28 days
  The highest dose at which there is <33% Dose Limiting Toxicity rate in the first cycle of treatment in a minimum of 6 patients.
Determine the Recommended Phase 2 Dose (RP2D) of emavusertib monotherapy (Phase 1) | 24 months
  The RP2D will be determined by the Clinical Safety Committee (CSC) in consultation with the Sponsor, considering all aspects of safety, tolerability, biologic activity, pharmacokinetics and preliminary efficacy in the trial population. The intent of an RP2D is to provide a dose and schedule that will maximize the opportunity for clinical benefit, while minimizing the risk of toxicity.
Determine Maximum Tolerated Dose (MTD) of emavusertib in combination with venetoclax (Phase 1b) | 28 days
  The highest dose at which there is <33% Dose Limiting Toxicity rate in the first cycle of treatment in a minimum of 6 patients.
Determine the Recommended Phase 2 Dose (RP2D) of emavusertib in combination with venetoclax (Phase 1b) | 24 months
  The RP2D will be determined by the Clinical Safety Committee (CSC) in consultation with the Sponsor, considering all aspects of safety, tolerability, biologic activity, pharmacokinetics and preliminary efficacy in the trial population. The intent of an RP2D is to provide a dose and schedule that will maximize the opportunity for clinical benefit, while minimizing the risk of toxicity.
To assess anti-cancer activity (Phase 2a - AML patients) | 24 months
  Proportion of patients who achieve complete response (CR) + complete response with partial hematological recovery (CRh)
To assess anti-cancer activity (Phase 2a - hrMDS patients) | 24 months
  Overall response rate: proportion of patients who achieve CR+ partial response (PR)
To assess safety (Phase 1b) | 24 months
  Clinical safety assessments including frequency of adverse events (AEs)

SECONDARY OUTCOMES:
To characterize the pharmacokinetic (PK) parameters of emavusertib measured by maximum plasma concentration (Cmax) (Phase 1 and 1b) | 24 months
  maximum plasma concentration (Cmax)
To characterize the pharmacokinetic (PK) parameters of emavusertib measured by trough plasma concentration (Cmin) (Phase 1 and Phase 1b) | 24 months
  trough plasma concentration (Cmin)
To characterize the pharmacokinetic (PK) parameters of emavusertib measured by Time to maximum plasma concentration (Tmax) (Phase 1 and 1b) | 24 months
  Time to maximum plasma concentration
To characterize the pharmacokinetic (PK) parameters of emavusertib measured by Area under the plasma concentration versus time curve(AUC) [0-24] (Phase 1 and 1b) | 24 months
  Area under the plasma concentration-time curve from 0 to 24 hours
To characterize the pharmacokinetic (PK) parameters of emavusertib measured by Area under the plasma concentration-time curve from 0 to infinity (AUC[INF]) (Phase 1 and 1b) | 24 months
  Area under the plasma concentration-time curve from 0 to infinity
To characterize the pharmacokinetic (PK) parameters of emavusertib measured by Plasma terminal elimination half-life (T 1/2) (Phase 1 and 1b) | 24 months
  Plasma terminal elimination half-life (T 1/2)
To assess clinical response (Phase 1 and 1b) | 24 months
  For AML: assessed by proportion of patients who reach complete response (CR) + complete response with partial hematological recovery (CRh) assessed by proportion of patients who reach complete response with incomplete hematologic recovery (CRi) or CR or CRh For hrMDS: overall response rate of CR+partial response (PR)
To assess clinical response (Phase 1 and 1b) | 24 months
  Assessed by transfusion independence
To assess tolerability and long term safety (Phase 2a) | 24 months
  Clinical safety assessments including frequency of adverse events (AEs)
To assess clinical response (Phase 2a) | 24 months
  For AML - assessed by proportion of patients who achieve CR or CRh or CRi; For hrMDS - assessed by proportion of patients who achieve CR or PR or marrow complete response (mCR)
To assess clinical response (Phase 2a) | 24 months
  Assessed by duration of response (DOR)
To assess clinical response (Phase 2a) | 24 months
  Assessed by time to response
To assess clinical response (Phase 2a) | 24 months
  Assessed by transfusion independence
To assess clinical response (Phase 2a) | 24 months
  Assessed by overall survival (OS)

CONTACTS AND LOCATIONS:
Locations (32):
- United States (12):
  - Moffitt Cancer Center, Tampa, Florida
  - Winship Cancer Institute, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Oncology Hematology West, PC dba Nebraska Cancer Specialists, Omaha, Nebraska
  - University of Rochester Medical Center, Rochester, New York
  - Albert Einstein Medical College, The Bronx, New York
  - Novant Health Hematology - Forsyth, Winston-Salem, North Carolina
  - The Ohio State University Wexner Medical Center - James Cancer Hospital, Columbus, Ohio
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Vseobecna Fakultni nemocnice v Praze, Prague, Czechia
- France (3):
  - Service d'hématologie clinique CHU de Nice, Nice
  - APHP - Sorbonne Universite, Paris
  - APHP - Hopital Saint Louis, Paris
- Germany (5):
  - Marien Hospital Dusseldorf; Klinik fur Onkologie und Hamatologie, Palliativmedizin, Düsseldorf
  - Universitätsklinikum Hamburg-Eppendorf (UKE), Hamburg
  - Universitatsklinikum Leipzig; Medizinische Klinik und Poliklinik I, Leipzig
  - Klinikum rechts der Isar der Technischen Universitat Munchen, München
  - Universitatsklinikum Munster, Münster
- Israel (3):
  - Soroka University MC, Beersheba
  - Edith Wolfson Medical Center, Holon
  - Hadassah University MC, Jerusalem
- Italy (2):
  - Azienda Ospedaliera Santa Croce e Carle, Cuneo
  - Instituto Romagnolo per lo Studio dei Tumori "Dino Amadori", Meldola
- Poland (2):
  - Uniwersyteckie Centrum Kliniczne Osrodek Badan Klinicznych Wczesnych Faz, Gdansk
  - University Hospital in Krakow, Krakow
- Spain (4):
  - Hospital de la Santa Creu I Sant Pau (Neuvo Hospital), Barcelona
  - Hospital Universitaro del a Princesa, Madrid
  - MD Anderson Cancer Center Madrid, Madrid
  - Hospital Universitario Virgen del Rocio, Seville

IPD SHARING:
Plan to Share IPD: No